CLINICAL TRIAL: NCT00307021
Title: Bridging Safety & Immunogenicity Study of GSK Biologicals' Candidate Malaria Vaccine RTS,S/AS01E (0.5 mL Dose) to RTS,S/AS02D (0.5 mL Dose) Administered IM According to a 0, 1, 2-Month Schedule in Gabonese Children Aged 18 Months to 4 Years
Brief Title: Double-blind Study of Safety and Immunogenicity of Two Candidate Malaria Vaccines in Gabonese Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 105874
Record Dates: First submitted 2006-02-16; First posted 2006-03-27 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Malaria
Keywords: Parasitic Diseases; Malaria, Falciparum; Malaria; Coccidiosis
MeSH Terms: conditions — Malaria; Parasitic Diseases; Malaria, Falciparum; Coccidiosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Group A (Active Comparator)
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- Group B (Experimental)
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049

INTERVENTIONS:
Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049 — 3-dose intramuscular injection, 2 different formulations

SUMMARY:
GSK Biologicals is developing a number of candidate malaria vaccines for the routine immunization of infants and children living in malaria-endemic areas. The candidate vaccines are designed to offer protection against malaria disease due to the parasite Plasmodium falciparum. Candidate vaccines containing the RTS,S antigen would also provide protection against infection with hepatitis B virus (HBV). This study will evaluate two candidate vaccines. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* A male or female child between 18 months and 4 years of age (up to but not including 5th birthday) at the time of first vaccination.
* Written or oral, signed or thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. return for follow-up visits)

Exclusion criteria:

* Acute disease at the time of enrolment.
* Serious acute or chronic illness determined by clinical or physical examination and laboratory screening tests.
* Laboratory screening tests for haemoglobin, total white cell count, platelets, ALT and creatinine out of range.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s) with the exception of tetanus toxoid.
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins, blood transfusions or other blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Previous participation in any other malaria vaccine trial.
* Simultaneous participation in any other clinical trial.
* Same sex twin.
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2006-04-07; Primary Completion 2006-09-15 (Actual); Study Completion 2007-08-22 (Actual)

PRIMARY OUTCOMES:
Occurrence of SAEs. | From the time of first vaccination until one month post Dose 3
Antibody titers to the P. falciparum circumsporozoite repeat domain (anti-CS). | One month post Dose 3.

SECONDARY OUTCOMES:
Occurrence of solicited general and local reactions. | Over a 7-day follow-up period after each vaccination.
Occurrence of unsolicited symptoms. | After each vaccination over a 30-day follow-up
Anti-CS antibody titers. | Prior to vaccination, one month post Dose 2
Anti-Hepatitis B surface agent (anti-HBs) antibody titers. | Prior to vaccination, one month post Dose 2 and one month post Dose 3.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Agnandji ST, Fendel R, Mestre M, Janssens M, Vekemans J, Held J, Gnansounou F, Haertle S, von Glasenapp I, Oyakhirome S, Mewono L, Moris P, Lievens M, Demoitie MA, Dubois PM, Villafana T, Jongert E, Olivier A, Cohen J, Esen M, Kremsner PG, Lell B, Mordmuller B. Induction of Plasmodium falciparum-specific CD4+ T cells and memory B cells in Gabonese children vaccinated with RTS,S/AS01(E) and RTS,S/AS02(D). PLoS One. 2011 Apr 11;6(4):e18559. doi: 10.1371/journal.pone.0018559. PMID 21494604
- [Background] Lell B, Agnandji S, von Glasenapp I, Haertle S, Oyakhiromen S, Issifou S, Vekemans J, Leach A, Lievens M, Dubois MC, Demoitie MA, Carter T, Villafana T, Ballou WR, Cohen J, Kremsner PG. A randomized trial assessing the safety and immunogenicity of AS01 and AS02 adjuvanted RTS,S malaria vaccine candidates in children in Gabon. PLoS One. 2009 Oct 27;4(10):e7611. doi: 10.1371/journal.pone.0007611. PMID 19859560
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 105874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register